CLINICAL TRIAL: NCT06400797
Title: ESTimation of Outcome by Health-Care PRoviders Compared With TruE Outcome in Patients Undergoing Veno-arteriaL and Veno-venous ExtracorporeaL MembrAne Oxygenation
Brief Title: Estimation of Outcome and Quality of Life in ECMO Patients
Acronym: ESTRELLA
Status: Recruiting | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-RM-01
Record Dates: First submitted 2024-05-02; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Extracorporeal Membrane Oxygenation
Keywords: ECMO; health related quality of life; Outcome estimation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECMO patients: Patients recieving Venoarterial or Venovenous extracorporeal membrane oxygenation (VA-ECMO, VV-ECMO)
  Interventions: Other: estimation of patient outcome by health care providers

INTERVENTIONS:
Other: estimation of patient outcome by health care providers — On day 1 after study inclusion as well as day 4-7, the responsible health-care providers (at least one nurse, one resident and one consultant with the board certification intensive care medicine) will estimate the patient's expected functional outcome at 6 and 12 months after the start of ECMO therapy. Health-care providers responsible for the patient at that time will be surveyed (multiple questionnaires to detect specific differences within one person are not planned). For the purpose of functional outcome estimation, the modified Rankin scale (mRS) is used.

SUMMARY:
The availability as well as the use of extracorporeal membrane oxygenation (ECMO) systems for severe acute respiratory or cardiocirculatory failure is steadily increasing. The decision to initiate ECMO therapy is predominantly made in emergency situations, for which the focus is on acute survival. The decisions if a patient will profit from ECMO therapy are mainly made from clinical experience and educated guess by the attending team. However, it is unknown how useful these clinical predictions are. Therefore, this observational study will compare estimated and real outcome of ECMO patients.

DETAILED DESCRIPTION:
The availability as well as the use of extracorporeal membrane oxygenation (ECMO) systems for severe acute respiratory (veno-venous, vv-ECMO) or cardiocirculatory (veno-arterial, va-ECMO) failure is steadily increasing. Despite increasing experience of specialized centres, mortality of ECMO patients remains high and only about 50% survive the initial hospital stay. For those patients who do leave the hospital alive, quality of life after this invasive therapy with long stays in the intensive care unit (ICU) is often limited and participation in social life can be difficult. Quality of life and the life-impact after ECMO therapy is, in contrast to hard endpoints such as mortality, insufficiently studied and currently only scarce data exist from large prospective cohort studies. Further, predictive scores and associated risk factors for patient-centred outcomes are not available.

The decision to initiate ECMO therapy is predominantly made in emergency situations, for which the focus is on acute survival. As such, the long-term implications in terms of quality of life and life-impact of ECMO treatment enjoy only limited consideration at an early time point. Further, the existing scores for prediction in ECMO were developed for mortality and reliable data on long-term life-impact are scarce. Therefore, while these decisions are influenced by empirical factors like patient-age, point-of-care laboratory parameters (e.g. lactate) or the neurological status of the patient, the clinical experience and educated guess in terms of prognosis and potential treatment futility by the attending team remains a crucial factor. This applies not only to ECMO initiation but also to decisions on continuation and termination. This approach to decision-making may be problematic since it has been shown for other settings that clinicians tend to overestimate the success of an intervention. Currently, there are no data evaluating in how far this also applies to ECMO therapy and if indeed, there is a mismatch between estimated and observed outcomes in ECMO patients. Considering the crucial role of subjective prognosis estimates, it becomes of major interest to quantify the potential mis-calibration between clinicians estimated and observed outcomes. Further, factors like Outcome uncertainties, potential doubts regarding treatment utility vs futility, and the immediate finality of these demanding decisions expose ICU health-care personnel to a relevant psychological burden. As shown by Johnson-Coyle and colleagues, both moral distress and burnout have a negative impact on job satisfaction. Moral distress occurs when one believes to know what is ethically right but something or someone limits their ability to do the right thing. Preliminary studies have shown a high incidence of moral distress in the care of patients with mechanical circulatory support systems, with particularly pronounced stress among nursing personnel. If these factors have significant impact on professional judgement is not clear in this context.

In a small single centre pilot study, we prospectively recruited 50 va-ECMO patients at the University Hospital Duesseldorf from March until November 2023 and investigated if ECMO care providers could predict in-hospital mortality in these patients. For these 50 patients we obtained 135 completed questionnaires within 24 hours and 111 answered questionnaires at day 4 to7 after initiation of ECMO therapy from consultants, residents and nursing personnel. Out of 50 patients 21 patients (42%) died during the initial hospital stay. Overall sensitivity and specificity of estimates were 57.9% and 85.9% respectively at 24 hours after start of ECMO therapy (precision: 75%, accuracy: 74.1%, F1 score: 65.3%). In a subgroup analysis, consultants showed highest agreement of estimated and actual in hospital mortality, whereas residents showed lowest agreement (see table below). At day 4 to 7 overall predictions had lower sensitivity, accuracy, precision and F1-score as compared to estimates on day 1 after ECMO initiation, however specificity slightly increased (sens: 35% spec: 91.5% acc: 71.1% F1-score: 46.7% precision: 70%). Highest values for sensitivity, accuracy and F1-score, were reached in subgroup of nursing personnel (see table below). Notably, years of experience in critical care were higher in consultants and nursing personnel as compared to residents (consultants: 10.8 ± 6.7 years versus residents: 1.4 ± 1.5 years versus nursing personnel: 15.8 ± 10.4 years).

Based on the results of our pilot data, we hypothesize that:

1. Subjective prognosis estimates by health care providers underestimate (low sensitivity) actual mortality. We expect that this will also account for reduced functionality and quality of life.
2. Estimations will vary significantly between different groups of health care professionals and levels of experience in critical care as well as between different time points of assessment. Specifically we expect, that prediction accuracy will improve with higher years of experience in critical care and that predictions for mortality will be more accurate immediately after ECMO initiation as compared to later study time points. This might be influenced by the fact that a substantial number of patients with poor prognosis will die within the first four days of ECMO therapy. Hence, estimation of outcome in the remaining patients is more difficult.
3. Agreement between estimated and observed outcomes will differ significantly between centres with different levels of experience (high-volume versus low-volume centres). Expecting higher accuracy of outcome estimates in high-volume centres with higher experience as compared to low-volume centres.
4. Additionally, we expect that high levels of moral distress influence professional judgement leading to negative estimated prognosis and low precisions of estimations.

Therefore, we aim to conduct the ESTRELLA study as large nationwide multicentre prospective cohort study to dissect usability of clinical estimates for outcome prediction in ECMO patients and to identify suitable factors for prediction of poor functional health in these patients.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* start of ECMO therapy ≤24h
* written informed consent from patient or health-care proxy

Exclusion Criteria:

* age < 18 years
* Language barrier (communication in German/local language or English not possible).
* no ECMO therapy or ECMO therapy longer than 24h
* no written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients aged above 18 years in the ICU with a vv- or va-ECMO for less than 24 hours will be included.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Agreement between estimated outcome by healthcare providers and actual patient outcome on Modified Rankin scale mRS | 6 months and 12 months after ECMO therapy
  The primary endpoint of this study will be the agreement between functional performance of patients estimated by different healthcare provider groups and actual functional performance of patients after start of ECMO therapy measured by the 7-item mRS.

SECONDARY OUTCOMES:
Disability-free survival (WHODAS 2.0) | 6 months and 12 months after ECMO therapy
  As secondary endpoints we will assess disability free survival at 6 and 12 months after ECMO therapy using the WHODAS 2.0 questionnaire with a disability threshold of ≥16 % for mild disability and ≥35% for severe disability as described previously by Shulman et al.
Days alive and out of hospital (DAOH) | 6 months and 12 months after ECMO therapy
  we will assess Days alive and out of hospital at 6 and 12 months after initiation of ECMO therapy, as additional life impact parameter which was previously investigated in other cohorts
Moral distress | Day 1 and day 4-7 of ECMO therapy
  we will assess the level of moral distress of ICU health care providers (consultants, residents and nursing personnel) taking care of the individual patient using the Moral Distress Thermometer.

CONTACTS AND LOCATIONS:
Overall Officials: René M'Pembele, MD, Principal Investigator — Heinrich-Heine University, Duesseldorf; Sebastian Roth, MD, Principal Investigator — Heinrich-Heine University, Duesseldorf
Locations (1):
- University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.